CLINICAL TRIAL: NCT05537805
Title: Ultrasound Guided Transcervical Fallopian Tube Catheterization During Hysterosalpingo-foam Sonography in the Treatment of Proximal Tubal Obstruction
Brief Title: Ultrasound Guided Fallopian Tube Catheterization During Hysterosalpingo-foam Sonography (HyFoSy)
Acronym: HyFoSy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Yaakov Melcer, Prof, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0275-21-ASF
Record Dates: First submitted 2022-09-04; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-01

CONDITIONS: Fallopian Obstruction Tube
MeSH Terms: conditions — Fallopian Tube Diseases

STUDY DESIGN:
Intervention Model Description: Prospective cohort study in a tertiary referral center. Investigators evaluated the procedure on a group of 30 participants that were referred to our unit for proximal tubal occlusion demonstrated by hysterosalpingo-foam sonography or hysterosalpingography.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- proximal tubal occlusion (Experimental): Infertile patients that were referred to our unit for uni or bilateral proximal tubal occlusion demonstrated by HyFoSy or hysterosalpingography.
  Interventions: Procedure: Ultrasound guided transcervical fallopian tube catheterization during hysterosalpingo-foam sonography in the treatment of proximal tubal obstruction

INTERVENTIONS:
Procedure: Ultrasound guided transcervical fallopian tube catheterization during hysterosalpingo-foam sonography in the treatment of proximal tubal obstruction — The intervention included the usage of the modified cornual cannulation set (COOK) which was inserted through cervical canal to uterine cavity, followed by fallopian tube irrigation with contrast foam (Ex-EM) during hysterosalpingo-foam sonography under ultrasonographic imaging.

SUMMARY:
Investigate a novel ultrasound guided transcervical fallopian tube catheterization during hysterosalpingo-foam sonography in the treatment of proximal tubal obstruction.

DETAILED DESCRIPTION:
Tubal catheterization is usually reserved for infertility treatment in selected cases of proximal tubal occlusion. As the incidence of this condition is limited to approximately 10-20% of women with mechanical infertility, the hitherto published data concerning the best therapeutic approach for these patients is scarce.

Hysterolaparoscopy with dye instillation is considered the gold standard for comprehensive evaluation of the female reproductive organs. Moreover, while the gold standard for evaluation of the uterine cavity is diagnostic hysteroscopy and hydrosonography, tubal patency may be validated by either hystrosalpingography, or ultrasonic evaluation using Echovist-200. However, interpretation of the passage of contrast medium into the proximal portion of the tube remains somewhat uncertain.

Since hysterolaparoscopy with dye instillation, is an expensive and an invasive procedure, with potentially life-threatening risks, the search for a safer and less invasive techniques is still ongoing. In 2012, Hysterosalpingo-Foam Sonography was introduced as a new technique for assessing fallopian tube patency. During the exam, the passage of a hyper-echogenic foam composed of a mixture of gel and purified water can be visualized as it progresses from the uterine cavity through the fallopian tubes into the peritoneal cavity. Hysterosalpingo-foam sonography is a promising alternative for laparoscopy and hysterosalpingography with regard to accuracy and effectiveness and has been suggested as a first step test of tubal assessment since it is relatively safe, non (embryo-) toxic and non-invasive.

In the present report the investigators aim to perform an ultrasound guided transcervical fallopian tube catheterization during hysterosalpingo-foam sonographyin the treatment of proximal tubal obstruction. This "one stop - shop" procedure combines uterine cavity investigation and assessment of tubal patency, with the concomitant advantage of therapeutic tubal re-canalization.

ELIGIBILITY:
Inclusion Criteria:

• uni or/and bilateral proximal tubal occlusion.

Exclusion Criteria:

* ongoing pregnancy
* positive Human Chorionic Gonadotropin test
* active pelvic inflammatory disease
* vaginal bleeding
* presence of distal tubal occlusion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with proximal tubal obstruction who referred for tubal catheterization in order to achieve fallopian tube recanalization (patency). | 18 month
  Tubal patency after tubal catheterization procedure demonstrated by hysterosalpingo-foam sonography.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohi MP. Interventional Radiologist's Approach to Fallopian Tube Recanalization. Tech Vasc Interv Radiol. 2021 Mar;24(1):100736. doi: 10.1016/j.tvir.2021.100736. Epub 2021 Apr 16. PMID 34147190
- [Background] Wang JW, Rustia GM, Wood-Molo M, Tasse J, Tabriz D, Turba UC, Arslan B, Madassery S. Conception rates after fluoroscopy-guided fallopian tubal cannulation: an alternative to in vitro fertilization for patients with tubal occlusion. Ther Adv Reprod Health. 2020 Oct 8;14:2633494120954248. doi: 10.1177/2633494120954248. eCollection 2020 Jan-Dec. PMID 33103116
- [Background] Pyra K, Szmygin M, Dymara-Konopka W, Zych A, Sojka M, Jargiello T, Leszczynska-Gorzelak B. The pregnancy rate of infertile patients with proximal tubal obstruction 12 months following selective salpingography and tubal catheterization. Eur J Obstet Gynecol Reprod Biol. 2020 Nov;254:164-169. doi: 10.1016/j.ejogrb.2020.08.008. Epub 2020 Sep 16. PMID 32979628
- [Background] De Silva PM, Chu JJ, Gallos ID, Vidyasagar AT, Robinson L, Coomarasamy A. Fallopian tube catheterization in the treatment of proximal tubal obstruction: a systematic review and meta-analysis. Hum Reprod. 2017 Apr 1;32(4):836-852. doi: 10.1093/humrep/dex022. PMID 28184438